CLINICAL TRIAL: NCT02123485
Title: The Antidepressant Efficacy of Repetitive Transcranial Magnetic Stimulation ( rTMS) as add-on to Electroconvulsive Therapy (ECT). A Double Blind Randomized Controlled Trial.
Brief Title: The Antidepressive Effect of rTMS as add-on to ECT
Acronym: TMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruiting of patients difficult combined by lack of money
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Poul Erik Buchholtz, MD, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1-10-72-509-12
Record Dates: First submitted 2014-03-13; First posted 2014-04-25 (Estimated); Results first posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Depression
Keywords: Depression,; ECT,; rTMS,; Right prefrontal,; antidepressive efficacy
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low frequency rTMS (Experimental): Right prefrontal Low frequency (1 hz) repetitive transcranial magnetic stimulation, administered with 2 sessions each week
  Interventions: Device: Low frequency (1 hz) rTMS, as add-on to ECT
- Sham-rTMS (Sham Comparator): Sham right prefrontal rTMS 2 times a week
  Interventions: Device: Sham-rTMS

INTERVENTIONS:
Device: Low frequency (1 hz) rTMS, as add-on to ECT — Right prefrontal Low frequency (1 hz) repetitive transcranial magnetic stimulation as add-on to ECT.
  Arms: low frequency rTMS
Device: Sham-rTMS — Right prefrontal Low frequency (1 hz) sham-stimulation using af double blind placebo coil as add-on to ECT.
  Arms: Sham-rTMS

SUMMARY:
The aim of the present study is to investigate in which degree low frequency right prefrontal rTMS used ad add-on may potentiate the antidepressant effect of unilateral ECT and accelerate remission .

To investigate the correlation between blood concentration of specific inflammation makers and change in depressive symptoms during treatment

DETAILED DESCRIPTION:
ECT is a well-established and effective method for the treatment of severe depression. During the last decades, rTMS has appeared as a potential new non-invasive antidepressant method, which may be a potential alternative to ECT due to fewer side effects.

Both methods expose the brain to an electric current. But while ECT is associated with global cerebral stimulation elicited by an epileptic seizure, rTMS implies non-convulsive focal stimulation through a time varying magnetic field. Thus, the antidepressant effect of rTMS does not depend on seizure activity and consequently requires no anesthesia. In addition, rTMS seems not to be associated with cognitive disturbances.

Previous research indicates that the antidepressant effect of rTMS is associated with specific stimulation of the dorsolateral prefrontal cortex. The majority of clinically controlled studies have used high frequency stimulation of the left frontal cortex (1-4). Few have used right prefrontal low frequency rTMS, which has less side effects, such as local discomfort and a lower risk of releasing epileptic seizures, than high frequency stimulation (5-10). Both models have been used with varying results. Meta-analysis of the antidepressant effect of rTMS (11,x) have found a modest, statistically significant antidepressant effect but generally definite conclusions on the antidepressant effect of rTMS has been difficult to draw, probably because of small and selected study populations, varying ways of stimulation and other confounding factors in the clinical setting.

The important clinical question of whether rTMS may substitute ECT in the treatment of depression has almost exclusively been elucidated in studies using high frequency stimulation of the left frontal cortex. Some of these suggest that the effectiveness of rTMS is equal to that of ECT in non-delusional patients (12-19). However, a recent investigation has compared the antidepressant efficacy and side effects of right prefrontal low frequency rTMS with ECT. In this study the mean Hamilton total 17-item (HAM-D score) scores were reduced significantly over time in both groups (ECT: p<0.001, rTMS: p<0.001); but ECT was more effective than rTMS on a short term after 3 weeks of treatment. The outcome did not point to right frontal low frequency rTMS as a first line substitute for ECT, but it might have place in the treatment of depression as add on to other types of treatment.

ECT is normally administered 3 times a week for 3-4 weeks. Daily treatment sessions might accelerate remission, but is impossible because of cognitive side effects. However, rTMS seems not to be associated with reduction in cognitive performance and might potentiate the antidepressant efficacy of ECT. Therefore the investigators have found it clinical interesting to investigate in which degree low frequency right prefrontal rTMS used ad add-on may potentiate the antidepressant effect of unilateral ECT and accelerate remission .

In addition we want to investigate te correlation between change in depressive symptoms and

-blood concentration of specific inflammation CNS- makers

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to the Psychiatric Hospital of Aarhus

* Patients referred for ECT
* Age 18-80 years
* Moderate or severely depressed patients (ICD-10(DSM-IV)
* HAM-D score (17-item) ≥20 and/or Ham-D subscale ≥10.

Exclusion Criteria:

* Organic brain disease
* Epilepsy or disposition to epilepsy
* Metallic objects in chest or brain
* Cardiac pacemaker
* Somatic diseases associated with brain dysfunction
* Pregnancy
* Severe agitation or delirium
* Alcohol or drug dependence (ICD-10)
* Use of coercive measures
* The patient does not wish to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Poul Erik Buchholtz, MD, Principal Investigator — Poul Erik Buchholtz, MD Telephone: 004578472109 Email: poulhans@rm.dk
Locations (1):
- Aarhus University Hospital, Risskov, Aarhus, Risskov, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Right Prefrontal Low Frequency (1 hz) Repetitive Transcranial Magnetic Stimulation (rTMS): Right prefrontal Low frequency (1 hz) repetitive transcranial magnetic stimulation, administered with 2 sessions each week
  Low frequency (1 hz) rTMS, as add-on to ECT: Right prefrontal Low frequency (1 hz) repetitive transcranial magnetic stimulation as add-on to ECT.
- Sham- Right Prefrontal Low Frequency (1 hz) Repetitive Transcranial Magnetic Stimulation (rTMS): Sham right prefrontal rTMS 2 times a week
  Sham-rTMS: Right prefrontal Low frequency (1 hz) sham-stimulation using af double blind placebo coil as add-on to ECT.
Period: Overall Study
Arm/Group | Right Prefrontal Low Frequency (1 hz) Repetitive Transcranial Magnetic Stimulation (rTMS) | Sham- Right Prefrontal Low Frequency (1 hz) Repetitive Transcranial Magnetic Stimulation (rTMS)
Started | 18 | 17
Completed | 17 | 17
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low Frequency Repetitive Transcranial Magnetic Stimulation (rTMS): Right prefrontal Low frequency (1 hz) repetitive transcranial magnetic stimulation, administered with 2 sessions each week
  Low frequency (1 hz) rTMS, as add-on to ECT: Right prefrontal Low frequency (1 hz) repetitive transcranial magnetic stimulation as add-on to ECT.
- Total: Total of all reporting groups
Arm/Group | Low Frequency Repetitive Transcranial Magnetic Stimulation (rTMS) | Sham-rTMS | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Full Range); unit: years] | 50 [19 to 80] | 47 [21 to 79] | 49 [19 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 5 | 5 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 18 | 17 | 35
Hamilton depression scale score [Mean (Full Range); unit: units on a scale] — The Hamilton (17 -item) Rating Scale for Depression is a clinician-administered assessement scale, that contains 17 items pertaining to symptoms of depression experienced over the past week. Full range = 0-52.
  The Hamilton 6-item subscale coveres 6 core symptoms of the 17 items. Full range = 0-22
  The major depression inventory scale is a self-reported modd questionnaire which is able to generate an estimate of symptom severety. The scale coveres 10 items. Full range =0-50 Increasing scores correlate to increasing severity of depression on all of the above mentioned scores.
  units on a scale
    Hamilton depression rating scale (17-item) | 24 [14 to 30] | 26 [19 to 37] | 25 [14 to 37]
    Hamilton depression rating scale (6-item) | 13 [8 to 16] | 13 [10 to 17] | 13 [8 to 17]
    Major Depression inventory | 45 [31 to 50] | 41 [30 to 50] | 43 [30 to 50]
Number of patients with Severe depression [Count of Participants; unit: Participants] | 15 | 17 | 32
number of patients with bipolar depressive [Count of Participants; unit: Participants] | 1 | 6 | 7
number of patients with melancholic depression [Count of Participants; unit: Participants] | 16 | 13 | 29
number of patients with psychotic depression [Count of Participants; unit: Participants] | 2 | 3 | 5
Antidepressant drug treatment [Count of Participants; unit: Participants] | 18 | 16 | 34

OUTCOME MEASURES:

1. Primary Outcome: Remission
Description: The Hamilton (17 -item) Rating Scale for Depression is a clinician-administered assessement scale, that contains 17 items pertaining to symptoms of depression experienced over the past week. The total range is 0-52.Higher scores mean a worse outcomeRemission is defined by a Hamilton 17-item total score < 8.
Time Frame: 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Low Frequency rTMS | Sham-rTMS
Number analyzed (Participants) | 17 | 17
Participants | 7 | 10
Statistical Analysis 1: Comparison: Low Frequency rTMS vs Sham-rTMS; Test type: Superiority; p = 0.30, Chi-squared

2. Secondary Outcome: Response
Description: The Hamilton (17 -item) Rating Scale for Depression is a clinician-administered assessement scale, that contains 17 items pertaining to symptoms of depression experienced over the past week. The total range is 0-52.Higher scores mean a worse outcome. Response is defined by a reduction in the Hamilton 17 item score of >= 50%
Time Frame: 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Low Frequency rTMS | Sham-rTMS
Number analyzed (Participants) | 17 | 17
Participants | 11 | 13

ADVERSE EVENTS:
Time Frame: 7 weeks
Description: All-Cause Mortality monitored/assessed in all participants who completed the study. Serious and Other adverse events were monitored/assessed in 26 participants (74% of the population).
Arm/Group | Low Frequency rTMS | Sham-rTMS
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/14
Other Adverse Events (participants affected / at risk) | 4/12 | 3/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Frequency rTMS (N=12) | Sham-rTMS (N=14)
severe confusion (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Frequency rTMS (N=12) | Sham-rTMS (N=14)
mild discomfort during treatment (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
mild headache (Nervous system disorders) | 4 (6) | 3 (4)

LIMITATIONS AND CAVEATS:
The study is under-powered

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT02123485/Prot_SAP_000.pdf